CLINICAL TRIAL: NCT05817838
Title: Testing a Multilevel, Multicomponent, Multigenerational Dietary Intervention to Improve Southeast Asian Children's Diets
Brief Title: Using Family-Based Approaches to Improve Healthy Eating for Southeast Asian Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Connecticut (Other); Center for Southeast Asians (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022003499; 1R01DK128197-01A1 (NIH)
Record Dates: First submitted 2023-03-21; First posted 2023-04-18 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-12

CONDITIONS: Diet, Healthy
Keywords: Asian Americans; Cambodian Americans; Hmong Americans; Vietnamese Americans; Laotian Americans; child; parents

STUDY DESIGN:
Intervention Model Description: Adult-child pairs will be randomized to: (1) financial incentive only arm that will receive weekly $15 financial incentive coupons to subsidize purchase of healthy foods at a local SEA grocery store; or (2) financial incentive plus twice-monthly, family-based group nutrition education at the Center for SEA led by SEA community health workers; three motivational interviewing (MI) calls by trained community health workers; dietary norms messaging for adults (via weekly text messages) and for children (via Infographics at nutrition education sessions); and weekly $15 financial incentive coupons to subsidize purchase of healthy foods at SEA grocery stores; or (3) an Academic Engagement attention control arm that will follow the structure of the financial incentive plus nutrition education, MI and text messages and infographics arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Attention control: Academic Engagement (Other): This intervention will be delivered using a similar format and schedule as the financial incentive+nutrition education, motivational interviewing and dietary norms intervention group (i.e., 11 community health worker led in-person group based sessions at the Center for Southeast Asians, 3 MI phone calls, and text messages). The content will focus on family-specific family engagement methods to improve children's academic outcomes.
  Interventions: Other: School Engagement
- Financial incentive only (Experimental): Participants will receive weekly financial incentive coupons to purchase eligible foods at the partnering Southeast Asian grocery store. Research Assistants will explain the coupon procedures during the randomization phone call. Research Assistants will mail the adult a schedule of coupon disbursement dates. RAs will mail one month's worth of coupons (4, $15 coupons) to each adult's home. Coupons will be used at point-of-sale. Participants' will receive an automated weekly text message via Qualtrics directing them to upload their photos to the system if they used coupons during that week.
  Interventions: Behavioral: Financial Incentives
- Financial incentive + nutrition education, motivational interviewing, dietary norms messages (Experimental): The intervention consists of a) four $15 financial incentive coupons each month; b) twice-monthly group-based nutrition education at the Center for SEA; c) motivational interviewing (months 1, 3, 5); and d) weekly dietary norms text messages sent to adults and twice-monthly dietary norms infographics presented at nutrition education sessions for children. The research assistants will disburse one months' worth of the financial incentive coupon at the nutrition education sessions (or home mailings for absent participants). Families will attend 11 fortnightly, group-based nutrition education sessions lasting one hour. Southeast Asian community health workers will lead the sessions. Research assistants trained in motivational interviewing will call the adults. The calls will last 15-20 minutes. Adults will receive a series of weekly, interactive descriptive dietary norms text messages. Children will see descriptive dietary norms infographics at children's nutrition education sessions.
  Interventions: Behavioral: Financial Incentives and Multilevel Multicomponent

INTERVENTIONS:
Behavioral: Financial Incentives — For six months, families will receive weekly, $15 financial incentives to purchase healthy foods and beverages at a partnering Southeast Asian grocery store
  Arms: Financial incentive only
Behavioral: Financial Incentives and Multilevel Multicomponent — For six months, families will receive weekly, $15 financial incentives to purchase healthy foods and beverages at a partnering Southeast Asian grocer store, in-person, group-based nutrition education with other Southeast Asian families, text messages and motivational interviewing
  Arms: Financial incentive + nutrition education, motivational interviewing, dietary norms messages
Other: School Engagement — For six months, families will attend in-person, group-based school engagement education with other Southeast Asian families designed to improve youths' academic outcomes. Families will receive text messages and motivational interviews. At the end of the six months, families will receive the equivalent of the six months worth of weekly, $15 financial incentives.
  Arms: Attention control: Academic Engagement

SUMMARY:
This small scale healthy eating study provides Southeast Asian families with children ages 6 to 11 with a family-based nutrition education, one-on-one interviews to help with motivation to eat health, text messaging, and coupons to purchase health foods and beverages. Since this is a small scale study that is a pilot intervention, the main goal of this intervention is to determine if it is feasible, meaning, can it be done. The second goal of this intervention is to determine if there are meaningful improvements in children's healthy eating patterns, body mass index and HbA1c. The third goal is to see if the intervention improves parent's diet quality, HbA1c and the home food environment. These study findings will be used to determine whether a larger clinical trial is needed, and if so, how it should be done.

DETAILED DESCRIPTION:
This intervention reflects the investigative team's eight year and ongoing academic-community research partnership with the Center for Southeast Asians (SEA) in Rhode Island, formative work with SEA families, and the team's extensive experience conducting successful dietary interventions. The current study is a pilot feasibility study that tests an innovative multilevel, multicomponent, multigenerational dietary intervention to improve diet quality among SEA children.

75 SEA families with children ages 6 to 11 years will be recruited from Providence County, Rhode Island. Adult-child pairs will be randomized to: (1) financial incentive only arm that will receive weekly $15 financial incentive coupons to subsidize purchase of healthy foods at a local SEA grocery store; or (2) financial incentive plus twice-monthly, family-based group nutrition education at the Center for SEA led by SEA community health workers; three motivational interviewing (MI) calls by trained community health workers; dietary norms messaging for adults (via weekly text messages) and for children (via Infographics at nutrition education sessions); and weekly $15 financial incentive coupons to subsidize purchase of healthy foods at SEA grocery stores; or (3) an Academic Engagement attention control arm that will follow the structure of the financial incentive plus nutrition education, MI and text messages and infographics arm. The primary outcomes are study feasibility and clinically meaningful improvement in child's diet quality (measured by healthy eating index). Secondary outcomes are clinically meaningful changes in children's body mass (~ 2kg weight loss or no weight gain), HbA1c (0.5%) and parent's diet quality, HbA1c and the home food environment. These study findings will be used to inform a future, larger clinical trial.

ELIGIBILITY:
Inclusion Criteria for Adults:

* Hmong, Cambodian, Laotian or Vietnamese
* the child's parent, legal guardian or grandparent
* live with the child
* age 18 or older
* knowledgeable about the child's diet
* responsible for household food preparation
* read/speak English, Hmong, Khmer, Vietnamese and/or Lao
* own a smartphone
* be willing to shop at the partner SEA grocery store

Exclusion Criteria for Adults:

* participation in weight-related studies in the past 12 months
* medical conditions that would affect participation (e.g., hospitalization due to type 2 diabetes in past year)

Inclusion Criteria for Children:

* Hmong, Cambodian, Laotian or Vietnamese
* age 6 to 11 years
* read/speak English
* Veggie Meter score ≤400

Exclusion Criteria for Children:

* disabilities that would affect participation
* chronic conditions affecting growth or diet
* medications affecting weight or metabolism

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Study Methods As Assessed by Rate of Participant Enrollment Each Month | Study enrollment to six-month follow-up
  Feasibility will be demonstrated if 7 enrolled Southeast Asian families per month are recruited on average over 12 months
Feasibility of Study Methods As Assessed by Participant Retention at 6-Months Study Completion | Study enrollment to six-month follow-up
  Feasibility will be demonstrated if 80% of enrolled families are retained at 6 months
Feasibility of Study Methods As Assessed by Participant Attendance at Group Sessions at 6-Months Study Completion | Study enrollment to six-month follow-up
  Feasibility will be demonstrated if 0% of enrolled families attend in-person sessions
Acceptability of the Intervention As Assessed by Participant Favorability Rating of the Intervention at Six-Months | Study enrollment to six-month follow-up
  Acceptability for each intervention component will be achieved if at least 70% of participants rate the component as "favorable" or "very favorable" on the measure of acceptability

SECONDARY OUTCOMES:
Diet quality as Assessed by 24-Hour Dietary Recall - Child | Study enrollment to six-month follow-up
  24-Hour dietary recall data will be converted to Healthy Eating Index scores to provide overall and subcomponent scores.
Fruit and vegetable intake as Assessed by The Veggie Meter - Child | Study enrollment to six-month follow-up
  Children's fruit and vegetable intake will be determined using the Veggie Meter, which is an objective measure of dermal carotenoids over a two month period.
Height ( Meters) as Assessed by Portable Stadiometer - Child and Adult | Study enrollment to six-month follow-up
  Objectively assessed height will be measured by research assistants using a portable stadiometer.
Weight (Kilograms) as Assessed by Tanita Body Scale - Child and Adult | Study enrollment to six-month follow-up
  Objectively assessed weight will be measured by research assistants using the Tanita Body Weight Scale.
Body Mass Index (BMI) as Assessed by the Ratio of Height/Weight (kg/m^2) - Child and Adult | Study enrollment to six-month follow-up
  Weight and height measures will be combined to compute Body Mass Index. Body Mass Index will be determined using appropriate child and adult reference values, respectively.
Waist Circumference (Inches) as Assessed by Seca Flexible Tape Measure - Child and Adult | Study enrollment to six-month follow-up
  Objectively assessed waist circumference will be measured by research assistants. Waist circumference categories will be determined using appropriate child and adult reference values, respectively.
Height (Feet and Inches) as Assessed by Portable Stadiometer - Child and Adult | Study enrollment to six-month follow-up
  Objectively assessed height, weight and waist circumference will be measured by research assistants. Body Mass Index and waist circumference categories will be determined using appropriate child and adult reference values, respectively.
Beverage Intake as Assessed by the Beverage Intake Questionnaire (Ounces) - Adult | Study enrollment to six-month follow-up
  Adult participants will complete a brief questionnaire to measure beverage intake (BEVQ-15).
Food Behaviors as Assessed by the Townsend Food Behaviors Checklist (units on a scale) - Adult | Study enrollment to six-month follow-up
  Adult participants will complete the Townsend Food Behaviors Checklist regarding consumption of foods and healthy food-related behaviors.
Fruit and Vegetable Intake as Assessed by The Veggie Meter Score | Study enrollment to six-month follow-up
  A Veggie Meter score (objective measure of fruit and vegetable intake) will be obtained for adults.
Home Food Environment as Assessed by a Food Inventory Checklist (units on a scale) | Study enrollment to six-month follow-up
  Adults will complete a self-report survey of the home food environment using the 23-item Home Food Inventory checklist.
HbA1c - adult and child | Study enrollment to six-month follow-up
  Child and adult HbA1c trained research staff will conduct finger sticks using established protocols (detailed protocol in Protection of Human Subjects)

CONTACTS AND LOCATIONS:
Overall Officials: Akilah Dulin, PhD, Principal Investigator — Brown University; Kim Gans, PhD, MPH, LDN, Principal Investigator — University of Connecticut
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to outside individuals because the data obtained from this feasibility R01 will be used to inform a larger, fully-powered R01-equivalent clinical trial.